CLINICAL TRIAL: NCT03310268
Title: A Randomized, 8 Week Clinical Study to Evaluate the Efficacy of an Experimental Stannous Fluoride Dentifrice in the Relief of Dentinal Hypersensitivity
Brief Title: A Clinical Study to Evaluate a Stannous Fluoride Toothpaste for the Relief of Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 208153
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Results first posted 2019-05-20 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tin Fluorides; Sodium Fluoride; fluorophosphate; stannous chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Product (Experimental): Participants will be instructed to self administer experimental dentifrice containing 0.454% SnF2 and 0.072% sodium fluoride (NaF) (1450 parts per million [ppm] fluoride in total).
  Interventions: Other: 0.454% Stannous fluoride (SnF2) and 0.072% sodium fluoride (NaF): 1450 ppm fluoride in total
- Negative Control (Active Comparator): Participants will be instructed to self administer negative control dentifrice containing 1400 ppm fluoride as sodium monofluorophosphate (SMFP).
  Interventions: Other: 1400 ppm fluoride as sodium monofluorophosphate (SMFP)
- Positive Control (Active Comparator): Participants will be instructed to self administer positive control dentifrice containing SnCl2 and 0.15% NaF (1450 ppm fluoride in total).
  Interventions: Other: Stannous Chloride (SnCl2) and 0.15% NaF: 1450 ppm fluoride in total

INTERVENTIONS:
Other: 0.454% Stannous fluoride (SnF2) and 0.072% sodium fluoride (NaF): 1450 ppm fluoride in total — Participants will be instructed to apply experimental dentifrice (containing 454% SnF2 and 0.072% NaF, 1450 ppm fluoride in total), covering the full length of toothbrush head (full ribbon) and will brush twice daily (morning and evening) for one timed minute (in their usual manner) and expectorate.
  Arms: Test Product
Other: 1400 ppm fluoride as sodium monofluorophosphate (SMFP) — Participants will be instructed to apply negative control dentifrice (containing 1400 ppm fluoride as SMFP), covering the full length of toothbrush head (full ribbon) and will brush twice daily (morning and evening) for one timed minute (in their usual manner) and expectorate.
  Arms: Negative Control
Other: Stannous Chloride (SnCl2) and 0.15% NaF: 1450 ppm fluoride in total — Participants will be instructed to apply positive control dentifrice (containing SnCl2 and 0.15% NaF, 1450 ppm fluoride in total), covering the full length of toothbrush head (full ribbon) and will brush twice daily (morning and evening) for one timed minute (in their usual manner) and expectorate.
  Arms: Positive Control

SUMMARY:
The purpose of this study is to provide evidence of clinical efficacy of an experimental dentifrice containing stannous fluoride (SnF2) compared to regular fluoride dentifrice in the reduction of dentinal hypersensitivity (DH). This study will be considered successful if there is a statistically significant difference in the primary efficacy variable, change from baseline in Schiff sensitivity score, after 8 weeks of treatment.

DETAILED DESCRIPTION:
This will be a single centre, randomized, controlled, examiner-blind, 3 treatment arm, parallel group design study, stratified by maximum baseline Schiff sensitivity score (of the two selected test teeth), with a treatment period of 8 weeks. DH will be assessed following an acclimatization period of 2-6 weeks at Baseline, and after 4 and 8 weeks treatment. The study will be conducted in healthy participants with pre-existing self-reported and clinically diagnosed tooth sensitivity at Screening. A standard fluoride dentifrice with no specific anti-sensitivity, anti-gingivitis and anti-plaque activity will be included as the negative control. A Chinese marketed positive control dentifrice with sensitivity benefits (containing stannous chloride (SnCl2)) will also be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent indicating the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Male and female participants who, at the time of screening, are between the ages of 18 and 70 years, inclusive.
* Participants who are willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* Good general and mental health, in the opinion of the investigator or medically qualified designee.
* Male participants able to father children and female participants of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 5 days after the last dose of assigned treatment. Female subjects who are not of childbearing potential must these meet requirements: Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle-stimulating hormone (FSH) level confirming the post-menopausal state; have undergone a documented hysterectomy and/or bilateral oophorectomy; have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations) will be considered to be of childbearing potential.
* The following oral and dental inclusions will apply at Screening (Visit 1): Self-reported history of dentinal hypersensitivity lasting more than six months but not more than 10 years, good general oral health, with a minimum of 20 natural teeth, minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, that meet all of the following criteria: signs of facial/cervical gingival recession and/or signs of erosion or abrasion (EAR), tooth with Modified Gingival Index (MGI) score =0 adjacent to the test area (exposed dentine) only and a clinical mobility of ≤1, tooth with signs of sensitivity measured by a qualifying tactile stimulus (Yeaple ≤20g) qualifying evaporative air assessment (Schiff sensitivity score >=2). The following dental inclusions will apply at Baseline (Visit 2): Minimum of two, non-adjacent accessible teeth (incisors, canines, pre-molars), with signs of sensitivity, measured by response to a qualifying tactile stimulus (Yeaple ≤20g) and evaporative air assessment (Schiff sensitivity score ≥2). The two selected test teeth must have also qualified at Screening for this criteria. The Investigator will select two Test Teeth from those which meet both the tactile threshold and Schiff sensitivity score criteria, in addition to meeting all other criteria. Test teeth should not be adjacent to each other and preferably in different quadrants.

Exclusion Criteria:

* Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are GSK employees directly involved in the conduct of the study.
* Participation in another clinical study (including cosmetic studies), or receipt of an investigational drug within 30 days prior to the Screening visit and/or during study participation.
* Participation in another tooth desensitizing treatment study within 8 weeks of the Screening visit.
* Acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Pregnant female participants. This will be confirmed verbally at Screening and confirmed by Urine pregnancy testing (carried out on all female participants of child bearing potential) at the Baseline visit.
* Breastfeeding female participants.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Recent history (within the last year) of alcohol or other substance abuse.
* Unwilling or unable to comply with the lifestyle guidelines described in this protocol.
* Participants who have previously been enrolled in this study.
* General oral and dental exclusions: Dental prophylaxis within 4 weeks of Screening, tongue or lip piercing or presence of dental implants, gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of Screening, scaling or root planning within 3 months of Screening, teeth bleaching within 8 weeks of Screening, use of an over-the-counter (OTC) desensitizing product (e.g. dentifrice) and/or professional desensitizing treatment within 8 weeks of Screening. participants will be required to bring their current oral care products to the site in order to verify the absence of known anti-sensitivity ingredients.
* Specific dental exclusions for test teeth: sensitive tooth not expected to respond to treatment with an over-the-counter dentifrice in the opinion of the investigator, tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine.
* Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of Screening.
* Concomitant Medication: Daily doses of medication/treatments or traditional herbal ingredients/treatments which, in the opinion of the investigator, could interfere with the perception of pain. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, anti-depressants, mood-altering and anti-inflammatory drugs. Examples of herbal ingredients/treatments include clove oil, olive oil, or other treatments that are directly applied to the oral cavity for the treatment of oral health conditions. Currently taking antibiotics or has taken antibiotics within 2 weeks of Screening and/or Baseline, Daily dose of a medication which, in the opinion of the investigator, is causing xerostomia, Individuals who require antibiotic prophylaxis for dental procedures.
* Any participant who, in the judgment of the investigator, should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2017-11-18 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20739

REFERENCES:
- [Result] Tao D, Ling MR, Feng XP, Gallob J, Souverain A, Yang W, Alavi A. Efficacy of an anhydrous stannous fluoride toothpaste for relief of dentine hypersensitivity: A randomized clinical study. J Clin Periodontol. 2020 Aug;47(8):962-969. doi: 10.1111/jcpe.13305. Epub 2020 Jun 8. PMID 32391584
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=208153&attachmentIdentifier=1a806d67-323f-4822-b3cc-92adba3f227a&fileName=gsk-208153-protocol-redact.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=208153&attachmentIdentifier=2484f32d-d8f8-4e4d-8141-4adf6d0700fd&fileName=gsk-208153-reporting-and-analysis-plan-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in China.
Pre-assignment Details: A total of 688 participates were screened, out of which 185 participants were randomized in the study and 503 participants were not randomized as 474 participants did not meet study criteria, 6 were reported with adverse events, 3 because of protocol violation, 4 withdrew consent, and 3 because of unspecified reasons.
Groups:
- Test Product (0.454% SnF2 and 0.072% NaF [1450 Ppm Fluoride]): Participants were instructed to self administer experimental dentifrice containing 0.454% stannous fluoride (SnF2) and 0.072% sodium fluoride (NaF) (1450 parts per million [ppm] fluoride in total) which covered the full length of toothbrush head (full ribbon) and brushed twice daily (morning and evening) for one timed minute (in their usual manner) and then expectorated.
- Negative Control (1400 Ppm Fluoride as SMFP): Participants were instructed to self administer negative control dentifrice containing 1400 ppm fluoride as sodium monofluorophosphate (SMFP)which covered the full length of toothbrush head (full ribbon) and brushed twice daily (morning and evening) for one timed minute (in their usual manner) and then expectorated.
- Positive Control (SnCl2 and 0.15% NaF [1450 Ppm Fluoride]): Participants were instructed to self administer positive control dentifrice containing stannous chloride (SnCl2) and 0.15% NaF (1450 ppm fluoride in total) which covered the full length of toothbrush head (full ribbon) and brushed twice daily (morning and evening) for one timed minute (in their usual manner) and then expectorated.
Period: Overall Study
Arm/Group | Test Product (0.454% SnF2 and 0.072% NaF [1450 Ppm Fluoride]) | Negative Control (1400 Ppm Fluoride as SMFP) | Positive Control (SnCl2 and 0.15% NaF [1450 Ppm Fluoride])
Started | 62 | 62 | 61
Completed | 61 | 57 | 61
Not Completed | 1 | 5 | 0
Not completed — (Not specified) | 1 | 5 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all randomized participants who received at least 1 dose of study treatment. This population was based on the treatment the subject actually received.
Groups:
- Test Product (0.454% SnF2 and 0.072% NaF [1450 Ppm Fluoride]): Participants were instructed to self administer experimental dentifrice containing 0.454% SnF2 and 0.072% NaF (1450 ppm fluoride in total) which covered the full length of toothbrush head (full ribbon) and brushed twice daily (morning and evening) for one timed minute (in their usual manner) and then expectorated.
- Negative Control (1400 Ppm Fluoride as SMFP): Participants were instructed to self administer negative control dentifrice containing 1400 ppm fluoride as SMFP which covered the full length of toothbrush head (full ribbon) and brushed twice daily (morning and evening) for one timed minute (in their usual manner) and then expectorated.
- Positive Control (SnCl2 and 0.15% NaF [1450 Ppm Fluoride]): Participants were instructed to self administer positive control dentifrice containing SnCl2 and 0.15% NaF (1450 ppm fluoride in total) which covered the full length of toothbrush head (full ribbon) and brushed twice daily (morning and evening) for one timed minute (in their usual manner) and then expectorated.
- Total: Total of all reporting groups
Arm/Group | Test Product (0.454% SnF2 and 0.072% NaF [1450 Ppm Fluoride]) | Negative Control (1400 Ppm Fluoride as SMFP) | Positive Control (SnCl2 and 0.15% NaF [1450 Ppm Fluoride]) | Total
Number analyzed (Participants) | 62 | 62 | 61 | 185
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.2 (10.83) | 40.3 (9.12) | 39.4 (9.95) | 39.9 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 47 | 59 | 161
  Male | 7 | 15 | 2 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 62 | 62 | 61 | 185
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 62 | 62 | 61 | 185
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Stratification n (%) [Count of Participants; unit: Participants]
  Maximum baseline Schiff score 2 | 44 | 44 | 43 | 131
  Maximum baseline Schiff score 3 | 18 | 18 | 18 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score After 8 Weeks of Treatment
Description: The examiner assessed the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale which was scored as follows - 0: Participant did not respond to air stimulation; 1: Participant responded to air stimulus but does not request discontinuation of stimulus; 2: Participant responded to air stimulus and requested discontinuation or moves from stimulus; 3: Participant responded to stimulus, considered stimulus to be painful, and requested discontinuation of the stimulus. A reduction in Schiff Sensitivity score will be indicative of an improvement in sensitivity.
Time Frame: Baseline, Week 8
Population: The Intent-to-treat (ITT) population included those participants who were randomized, received at least 1 dose of study treatment, and had at least 1 post baseline efficacy evaluation. This population was based on the treatment to which the subject was randomized. The primary population for assessment of efficacy was the ITT population.
Measure: Mean (Standard Deviation); unit: Score on Scale
Groups:
- Positive Control (SnCl2 and 0.15% NaF [1450 Ppm Fluoride]): Participants were instructed to self administer positive control dentifrice containing SnCl2 and 0.15% NaF (1450 ppm fluoride in total) which covered the full length of toothbrush head (full ribbon) and brushedtwice daily (morning and evening) for one timed minute (in their usual manner) and then expectorated.
Arm/Group | Test Product (0.454% SnF2 and 0.072% NaF [1450 Ppm Fluoride]) | Negative Control (1400 Ppm Fluoride as SMFP) | Positive Control (SnCl2 and 0.15% NaF [1450 Ppm Fluoride])
Number analyzed (Participants) | 62 | 60 | 61
Score on Scale
  Schiff score at baseline | 2.22 (0.369) | 2.23 (0.385) | 2.18 (0.303)
  Schiff score at Week 8 | 1.69 (0.449) | 1.50 (0.526) | 1.70 (0.572)
  Change from baseline in Schiff score at Week 8 | -0.53 (0.562) | -0.72 (0.567) | -0.48 (0.591)
Statistical Analysis 1: Comparison: Test Product (0.454% SnF2 and 0.072% NaF [1450 Ppm Fluoride]) vs Negative Control (1400 Ppm Fluoride as SMFP); Test type: Other; p = 0.0476, ANCOVA; From ANCOVA model with treatment as factor and baseline Schiff score as covariate; Difference of Least Square mean = 0.19, 95% CI 2-sided [0.002 to 0.374], Standard Error of Mean 0.094 — Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment
Statistical Analysis 2: Comparison: Test Product (0.454% SnF2 and 0.072% NaF [1450 Ppm Fluoride]) vs Positive Control (SnCl2 and 0.15% NaF [1450 Ppm Fluoride]); Test type: Other; p = 0.8411, ANCOVA; From ANCOVA model with treatment as factor and baseline Schiff score as covariate; Difference of Least Square mean = -0.02, 95% CI 2-sided [-0.202 to 0.164], Standard Error of Mean 0.093 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Negative Control (1400 Ppm Fluoride as SMFP) vs Positive Control (SnCl2 and 0.15% NaF [1450 Ppm Fluoride]); Test type: Other; p = 0.0298, ANCOVA; From ANCOVA model with treatment as factor and baseline Schiff score as covariate; Difference of Least Square mean = 0.21, 95% CI 2-sided [0.020 to 0.393], Standard Error of Mean 0.094 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Tactile Threshold After 8 Weeks of Treatment
Description: The examiner assessed the response to tactile sensitivity using a Yeaple probe which allowed the application of a known force to the dentin surface, starting at 10 grams (g) and rising in increments of 10g until the tactile threshold or maximum force was reached. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth. At baseline, the maximum force used was 20g; at all subsequent visits, it was 80g.
Time Frame: Week 8
Population: The ITT population included those participants who were randomized, received at least 1 dose of study treatment, and had at least 1 post baseline efficacy evaluation. This population was based on the treatment to which the subject was randomized. The primary population for assessment of efficacy was the ITT population.
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Test Product (0.454% SnF2 and 0.072% NaF [1450 Ppm Fluoride]) | Negative Control (1400 Ppm Fluoride as SMFP) | Positive Control (SnCl2 and 0.15% NaF [1450 Ppm Fluoride])
Number analyzed (Participants) | 62 | 60 | 61
Grams
  Tactile threshold at baseline | 11.13 (2.294) | 11.42 (2.272) | 11.80 (3.032)
  Tactile threshold at Week 8 | 28.52 (22.846) | 36.49 (29.124) | 33.93 (24.902)
  Change from baseline at Week 8 | 17.38 (22.631) | 25.00 (28.769) | 22.31 (24.229)
Statistical Analysis 1: Comparison: Test Product (0.454% SnF2 and 0.072% NaF [1450 Ppm Fluoride]) vs Negative Control (1400 Ppm Fluoride as SMFP); Test type: Other; p = 0.1232, ANCOVA; From ANCOVA model with treatment and baseline Schiff stratification as factors and baseline tactile threshold as a covariate; Difference of Least Square mean = -7.20, 95% CI 2-sided [-16.376 to 1.975], Standard Error of Mean 4.649 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Test Product (0.454% SnF2 and 0.072% NaF [1450 Ppm Fluoride]) vs Positive Control (SnCl2 and 0.15% NaF [1450 Ppm Fluoride]); Test type: Other; p = 0.3793, ANCOVA; [statistical method as in outcome 2, analysis 1]; Difference of Least Square mean = -4.04, 95% CI 2-sided [-13.099 to 5.011], Standard Error of Mean 4.588 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Negative Control (1400 Ppm Fluoride as SMFP) vs Positive Control (SnCl2 and 0.15% NaF [1450 Ppm Fluoride]); Test type: Other; p = 0.4979, ANCOVA; [statistical method as in outcome 2, analysis 1]; Difference of Least Square mean = -3.16, 95% CI 2-sided [-12.330 to 6.017], Standard Error of Mean 4.648 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From screening up to Week 8
Arm/Group | Test Product (0.454% SnF2 and 0.072% NaF [1450 Ppm Fluoride]) | Negative Control (1400 Ppm Fluoride as SMFP) | Positive Control (SnCl2 and 0.15% NaF [1450 Ppm Fluoride])
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62 | 0/61
Other Adverse Events (participants affected / at risk) | 7/62 | 3/62 | 4/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (0.454% SnF2 and 0.072% NaF [1450 Ppm Fluoride]) (N=62) | Negative Control (1400 Ppm Fluoride as SMFP) (N=62) | Positive Control (SnCl2 and 0.15% NaF [1450 Ppm Fluoride]) (N=61)
Lip Ulceration (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Non infective Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Oral Herpes (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Angular Chelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulpitis Dental (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT03310268/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT03310268/SAP_001.pdf